CLINICAL TRIAL: NCT02601547
Title: PET-based Evaluation of Chemotherapy-induced Brain Damage in Lymphoma Patients -Implication in the Evaluation of Neuro-cognitive Function Alteration (LYMCOTEP)
Brief Title: PET-based Evaluation of Chemotherapy-induced Brain Damage in Lymphoma
Acronym: LYMCOTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 09 154 02
Record Dates: First submitted 2015-09-29; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma
Keywords: Positron-Emission Tomography; chemotherapy-induced brain damage; neuro-cognitive function alteration
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): 1. PET-FDG brain imaging and NPT should be performed at T0 (within the 15 days before chemotherapy), at Tf (within 1 month after chemotherapy termination), T+12 (Tf+12 months: within the first month after one year of achievement of chemotherapy). Several PET parameters should be calculated: minimal Standard Uptake Value (SUV), maximum SUV, and mean SUV for each of 20 cortical and sub-cortical territories.
  2. NPT scores (3 values) should be correlated with the five better values on PET-FDG.
  3. Each patient will be monitored along a time period of 18 months.
  4. Duration of the study: one year to include the 15 patients with all the exams; 18 months follow-up for each; total of 30 months.
  Interventions: Device: PET-FDG brain imaging and NPT

INTERVENTIONS:
Device: PET-FDG brain imaging and NPT — PET-FDG brain imaging and NPT should be performed at T0, at Tf (within 1 month after chemotherapy termination), T+12. Several PET parameters should be calculated: minimal SUV (Standard Uptake Value), maximum SUV, and mean SUV for each of 20 cortical and sub-cortical territories.
  Other Names: 18F-Fluoro-Desoxy-Glucose brain imaging and NPT

SUMMARY:
Positron emission tomography (PET) with 18-fluoro-deoxy-glucose (PET-FDG) is emerging as a promising approach for detecting brain lesions in dementia, among which Alzheimer's disease has been the most widely studied.

DETAILED DESCRIPTION:
Alteration of neuro-cognitive function induced by chemotherapy has been extensively documented in breast carcinoma patients. These modifications consist in the decrease of memory, intellectual capacity, speed analysis, and represent a real limitation for patients, sometimes durable. Aggressive lymphomas (diffuse large B cell lymphomas/DLBCL) represent a common disease, the standard being Rituximab-Cyclophosphamide-Doxorubicine-Vincristine-Prednisone (RCHOP) regiment which contains, as for breast cancer patients, anthracyclines. However, very little is known about the incidence and severity of cognitive function alteration in these patients. The occurrence of such complications should also be facilitated because of frail cognitive states due to age and co-morbidity. Cognitive function alteration is usually measured by neuropsychological tests (NPT) which are easy to handle and sensitive, but could lack specificity, in the context of general degradation which is often observed in hematological patients.

Positron emission tomography with 18-fluoro-deoxy-glucose (PET-FDG) is emerging as a promising approach for detecting brain lesions in dementia, among which Alzheimer's disease has been the most widely studied. In our center, the investigators have already described glucidic hypometabolism in several brain territories associated with Alzheimer's disease and other dementia. Moreover, uptake quantification and topography are useful markers for determining the type of the disease and progression. PET-FDG received very little attention for the detection of chemotherapy-induced brain damages.

ELIGIBILITY:
Inclusion Criteria:

* histologically documented DLBCL
* previously untreated
* with International Prognostic Index (IPI) 0 or 1, or 2 without general state alteration (OMS≤2)
* submitted to RCHOP regimen (according to GELA's standard protocol)
* normal pre-treatment brain CT scan
* able to give informed consent
* speaking well French language
* benefiting from general medical insurance
* registered in the national listing of patients for biomedical research.

Exclusion Criteria:

* IPI > or =3
* medical history of another cancer, or psychiatric or pre-dementia disorder, or convulsion
* barbituric regular use which can't be stop
* human immunodeficiency virus (HIV) patients
* unstable diabetes mellitus
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change of Standard Uptake Value | 1 month after chemotherapy termination
Change of Standard Uptake Value | 12 months after one year of achievement of chemotherapy

SECONDARY OUTCOMES:
change of functional learning test (WAIS) | 1 month after chemotherapy termination
change of functional learning test (WAIS) | 12 months after one year of achievement of chemotherapy
change of depression scale | 1 month after chemotherapy termination
change of depression scale | 12 months after one year of achievement of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Anne Julian, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France